CLINICAL TRIAL: NCT00925054
Title: Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous (SC) Doses of rAvPAL-PEG in Subjects With PKU
Brief Title: Dose-Finding Study to Evaluate the Safety, Efficacy, & Tolerability of Multiple Doses of rAvPAL-PEG in Subjects With PKU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PAL-002
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Phenylketonuria
Keywords: PKU; PEG PAL; BioMarin
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- rAvPAL-PEG 0.001 mg/kg (Experimental): Subjects will start on rAvPAL-PEG 0.001 mg/kg
  Interventions: Drug: rAvPAL-PEG 0.001 mg/kg
- rAvPAL-PEG 0.003 mg/kg (Experimental): Subjects will start on rAvPAL-PEG 0.003 mg/kg
  Interventions: Drug: rAvPAL-PEG 0.003 mg/kg
- rAvPAL-PEG 0.01 mg/kg (Experimental): Subjects will start on rAvPAL-PEG 0.01 mg/kg
  Interventions: Drug: rAvPAL-PEG 0.01 mg/kg
- rAvPAL-PEG 0.03 mg/kg (Experimental): Subjects will start on rAvPAL-PEG 0.03 mg/kg
  Interventions: Drug: rAvPAL-PEG 0.03 mg/kg
- rAvPAL-PEG 0.1 mg/kg (Experimental): Subjects will start on rAvPAL-PEG 0.1 mg/kg
  Interventions: Drug: rAvPAL-PEG 0.1 mg/kg

INTERVENTIONS:
Drug: rAvPAL-PEG 0.001 mg/kg — In Part 1, the planned starting dose levels is 0.001 mg/kg
  Arms: rAvPAL-PEG 0.001 mg/kg
Drug: rAvPAL-PEG 0.003 mg/kg — In Part 1, the planned starting dose levels is 0.003 mg/kg
  Arms: rAvPAL-PEG 0.003 mg/kg
Drug: rAvPAL-PEG 0.01 mg/kg — In Part 1, the planned starting dose levels is 0.01 mg/kg
  Arms: rAvPAL-PEG 0.01 mg/kg
Drug: rAvPAL-PEG 0.03 mg/kg — In Part 1, the planned starting dose levels is 0.03 mg/kg
  Arms: rAvPAL-PEG 0.03 mg/kg
Drug: rAvPAL-PEG 0.1 mg/kg — In Part 1, the planned starting dose levels is 0.1 mg/kg
  Arms: rAvPAL-PEG 0.1 mg/kg

SUMMARY:
The purpose of this study is to evaluate whether weekly injections of phenylalanine ammonia lyase (rAvPAL-PEG) can reduce blood phenylalanine concentrations in PKU subjects and whether repeated administration is safe.

DETAILED DESCRIPTION:
This is a 2 part, Phase 2, open-label dose-finding study in approximately 35 subjects with PKU. Seven dose cohorts are planned, each consisting of 5 subjects. In Part 1, the planned starting dose levels are those tested in PAL 001 (0.001, 0.003, 0.01, 0.03, 0.1, 0.3, and 1.0 mg/kg), provided no dose limiting toxicity was observed in PAL 001. In Parts 1 and 2, study drug will be administered by clinic staff.

Subjects who completed participation in PAL 001 will receive priority to participate in PAL 002. rAvPAL PEG naïve subjects will be enrolled to fill any dose cohort vacancies resulting from subjects who did not complete PAL 001 or who chose not to continue into PAL 002. In addition, if the number of dose cohorts determined in PAL 001 is less than 7, additional naïve subjects may be added to the existing dose cohorts to provide a total of approximately 35 subjects entering Part 1 of PAL 002. Furthermore, if serial dosing of cohorts in Part 1 of PAL 002 is stopped, additional subjects (either naïve subjects or PAL 001 subjects) may be added to the existing cohorts so that total study enrollment is approximately 35 subjects. In any of these cases, additional subjects will be enrolled sequentially from lowest to highest dose cohort.

Diet will not be altered during the course of this study, except as necessary for safety.

Subjects will be evaluated for safety and for blood Phe concentrations throughout the study. Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.

A Data Monitoring Committee will monitor the study.

ELIGIBILITY:
Inclusion Criteria:

* For subjects who did not participate in PAL-001, diagnosis of PKU with both of the following: Current blood Phe concentration of ≥ 600 mmol/L at Screening and average blood Phe concentration of ≥ 600 µmol/L over the past 3 years, using available data.
* For subjects who did not participate in PAL-001, evidence that the subject is a non-responder to Kuvan® treatment (ie, 4 weeks of treatment with 20 mg/kg/day of Kuvan®, insufficient response per investigator determination, and treatment end date ≥ 14 days prior to Day 1 [ie, first dose]). Subjects who have had a previous response to Kuvan® treatment but are not currently taking Kuvan® because of noncompliance and have been off treatment for ≥ 6 months prior to Screening are eligible for participation.
* Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
* Between the ages of 16 and 55 years, inclusive.
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
* Maintained a stable diet with no significant modifications during the 4 weeks preceding the administration of study drug.
* In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.
* Willing and able to comply with study procedures.

Exclusion Criteria:

* Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug.
* Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 3 months prior to Screening and during study participation.
* A prior reaction that included systemic symptoms (eg, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG containing product. Subjects with a prior systemic reaction of generalized rash may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer.
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
* Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
* Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
* Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
* Creatinine > 1.5 times the upper limit of normal.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Gershman, MD, Study Director — BioMarin Pharmaceutical
Locations (11):
- United States (11):
  - The Children's Hospital, Aurora, Colorado
  - Emory Universty, Decatur, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Washington University Center for Applied Research Sciences, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Mount Sinai School of Medicine, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Utah Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burton BK, Longo N, Vockley J, Grange DK, Harding CO, Decker C, Li M, Lau K, Rosen O, Larimore K, Thomas J; PAL-002 and PAL-004 Investigators. Pegvaliase for the treatment of phenylketonuria: Results of the phase 2 dose-finding studies with long-term follow-up. Mol Genet Metab. 2020 Aug;130(4):239-246. doi: 10.1016/j.ymgme.2020.06.006. Epub 2020 Jun 16. PMID 32593547
- [Derived] Longo N, Harding CO, Burton BK, Grange DK, Vockley J, Wasserstein M, Rice GM, Dorenbaum A, Neuenburg JK, Musson DG, Gu Z, Sile S. Single-dose, subcutaneous recombinant phenylalanine ammonia lyase conjugated with polyethylene glycol in adult patients with phenylketonuria: an open-label, multicentre, phase 1 dose-escalation trial. Lancet. 2014 Jul 5;384(9937):37-44. doi: 10.1016/S0140-6736(13)61841-3. Epub 2014 Apr 14. PMID 24743000

RESULTS

PARTICIPANT FLOW:
Groups:
- Starting Dose=0.001 mg/kg: Subjects will start on rAvPAL-PEG 0.001 mg/kg
- Starting Dose=0.003 mg/kg: Subjects will start on rAvPAL-PEG 0.003 mg/kg
- Starting Dose=0.01 mg/kg: Subjects will start on rAvPAL-PEG 0.01 mg/kg
- Starting Dose=0.03 mg/kg: Subjects will start on rAvPAL-PEG 0.03 mg/kg
- Starting Dose=0.1 mg/kg: Subjects will start on rAvPAL-PEG 0.1 mg/kg
Period: Overall Study
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose=0.1 mg/kg
Started | 7 | 9 | 13 | 1 | 10
Completed | 7 | 8 | 12 | 0 | 10
Not Completed | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose=0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (3.45) | 29.2 (5.95) | 26.5 (5.65) | 22.0 | 25.2 (8.60) | 26.1 (6.35)
Age, Customized [Count of Participants; unit: Participants]
  < 18 years of age | 0 | 0 | 0 | 0 | 2 | 2
  > or = 18 years of age | 7 | 9 | 13 | 1 | 8 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 6 | 0 | 4 | 20
  Male | 4 | 2 | 7 | 1 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 9 | 13 | 1 | 9 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 9 | 12 | 1 | 9 | 38
  Other | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 9 | 13 | 1 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Blood Phenylalanine Concentrations
Time Frame: Baseline, Week 1/Day 5, Week 7, Week 16/Day 106
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: umol/L
Groups:
- Starting Dose=0.001 mg/kg: Subjects with starting Dose=0.001 mg/kg
- Starting Dose=0.003 mg/kg: Subjects with starting Dose=0.003 mg/kg
- Starting Dose=0.01 mg/kg: Subjects with starting Dose=0.01 mg/kg
- Starting Dose=0.03 mg/kg: Subjects with starting Dose=0.03 mg/kg
- Starting Dose =0.1 mg/kg: Subjects with starting Dose =0.1 mg/kg
- Total: All subjects with different starting dose combined
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose =0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
umol/L
  Baseline | 1382.7 (191.40) | 1336.1 (344.87) | 1290.5 (459.43) | 846.0 | 1310.3 (319.01) | 1310.8 (353.86)
  Week 1 Day 5: number analyzed (Participants) | 7 | 8 | 13 | 1 | 10 | 40
  Week 1 Day 5 | 1405.3 (190.87) | 1276.3 (410.22) | 1216.5 (434.53) | 682.0 | 863.7 (307.59) | 1158.5 (403.63)
  Week 7: number analyzed (Participants) | 7 | 9 | 13 | 1 | 8 | 40
  Week 7 | 1436.0 (274.08) | 1324.8 (304.64) | 1108.7 (510.74) | 1849.0 | 1321.6 (350.78) | 1284.5 (405.75)
  week 16 Day 106: number analyzed (Participants) | 7 | 8 | 13 | 0 | 7 | 40
  week 16 Day 106 | 1284.0 (221.73) | 1049.4 (378.00) | 1093.5 (445.02) |  | 930.7 (331.36) | 1088.5 (367.67)

2. Secondary Outcome: Study Drug Related Adverse Events
Time Frame: Screening, Weeks 1-22
Population: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration and have post-treatment safety information (laboratory values, vital signs, adverse events, 12-lead electrocardiogram, antibodies, and physical examinations).
Measure: Count of Participants; unit: Participants
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose =0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
Participants | 5 | 9 | 11 | 1 | 10 | 36

3. Secondary Outcome: Number of Participants With Positive PAL IgG Antibody
Description: Antibody against PAL (phenylalanine ammonia lyase) measured over time
Time Frame: Baseline, Week 12
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose =0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
Participants
  Baseline | 3 | 2 | 2 | 0 | 0 | 7
  Week 12: number analyzed (Participants) | 7 | 8 | 12 | 1 | 10 | 38
  Week 12 | 7 | 8 | 12 | 1 | 10 | 38

4. Secondary Outcome: Number of Participants With Positive PAL IgM Antibody
Description: Antibody positivity over time
Time Frame: Baseline, Week 12
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose =0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
Participants
  Baseline | 1 | 2 | 5 | 0 | 4 | 12
  Week 12: number analyzed (Participants) | 7 | 8 | 12 | 1 | 10 | 38
  Week 12 | 4 | 3 | 8 | 0 | 10 | 25

5. Secondary Outcome: Number of Participants With Positive PEG IgM Antibody
Description: Antibody positivity over time
Time Frame: Baseline, Week 16
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose =0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
Participants
  Baseline | 1 | 2 | 2 | 0 | 0 | 5
  Week 16: number analyzed (Participants) | 7 | 8 | 12 | 1 | 10 | 38
  Week 16 | 7 | 7 | 8 | 0 | 9 | 34

6. Secondary Outcome: Number of Participants With Positive PEG IgG Antibody
Description: Antibody positivity over time
Time Frame: Baseline, Week 16
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose =0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
Participants
  Baseline | 2 | 5 | 7 | 1 | 4 | 19
  Week 16: number analyzed (Participants) | 7 | 8 | 12 | 1 | 10 | 38
  Week 16 | 6 | 7 | 12 | 0 | 9 | 34

7. Secondary Outcome: Percentage of Participants With Positive Neutralizing Antibodies [NAb]
Description: Antibody positivity over time
Time Frame: Baseline, Week 12
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose =0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
Participants
  Baseline | 0 | 0 | 0 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 7 | 8 | 12 | 1 | 10 | 38
  Week 12 | 0 | 0 | 1 | 0 | 3 | 4

8. Secondary Outcome: Percentage of Participants With Positive PAL IgE Antibody
Description: Antibody positivity over time
Time Frame: Baselline, Week 12
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose =0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
Participants
  Baseline: number analyzed (Participants) | 7 | 9 | 13 | 1 | 9 | 39
  Baseline | 0 | 0 | 0 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 7 | 8 | 12 | 1 | 10 | 38
  Week 12 | 1 | 0 | 0 | 0 | 0 | 1

9. Secondary Outcome: Percentage of Participants With Positive Anti-PAL-PEG IgE Antibodies
Description: Antibody positivity over time
Time Frame: Baseline, Week 12
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose =0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
Participants
  Baseline: number analyzed (Participants) | 7 | 9 | 13 | 1 | 9 | 39
  Baseline | 0 | 0 | 0 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 7 | 8 | 12 | 1 | 10 | 38
  Week 12 | 0 | 0 | 0 | 0 | 0 | 0

10. Other Pre Specified Outcome: Trough Concentration of BMN 165
Description: Plasma concentrations of rAvPAL-PEG (BMN 165)
Time Frame: Baseline, Baseline/pre-dose, Week 7, and Week 16/Day 106
Population: The PK population will consist of all subjects who received any amount of study drug and have post-treatment plasma BMN 165 concentration measurements.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose =0.1 mg/kg | Total
Number analyzed (Participants) | 7 | 9 | 13 | 1 | 10 | 40
ng/mL
  Baseline: number analyzed (Participants) | 7 | 9 | 13 | 1 | 0 | 30
  Baseline | 0 (0) | 0 (0) | 0 (0) | 0 |  | 0 (0)
  Baseline, pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  Baseline, pre-dose |  |  |  |  | 1.6 (5.06) | 1.6 (5.06)
  Week 7: number analyzed (Participants) | 7 | 9 | 13 | 1 | 8 | 38
  Week 7 | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0)
  Week 16-Day 106: number analyzed (Participants) | 7 | 8 | 12 | 0 | 9 | 36
  Week 16-Day 106 | 7.8 (20.52) | 3.1 (8.70) | 6.0 (14.54) |  | 0 (0) | 4.2 (12.74)

ADVERSE EVENTS:
Time Frame: Screening- Week 22
Arm/Group | Starting Dose=0.001 mg/kg | Starting Dose=0.003 mg/kg | Starting Dose=0.01 mg/kg | Starting Dose=0.03 mg/kg | Starting Dose=0.1 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9 | 0/13 | 0/1 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9 | 1/13 | 0/1 | 1/10
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9 | 13/13 | 1/1 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Starting Dose=0.001 mg/kg (N=7) | Starting Dose=0.003 mg/kg (N=9) | Starting Dose=0.01 mg/kg (N=13) | Starting Dose=0.03 mg/kg (N=1) | Starting Dose=0.1 mg/kg (N=10)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Starting Dose=0.001 mg/kg (N=7) | Starting Dose=0.003 mg/kg (N=9) | Starting Dose=0.01 mg/kg (N=13) | Starting Dose=0.03 mg/kg (N=1) | Starting Dose=0.1 mg/kg (N=10)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (10) | 4 (5) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (7) | 2 (5) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 3 (3)
Injection site dermatitis (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (3) | 4 (8) | 4 (12) | 0 (0) | 4 (5)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 2 (6) | 1 (2) | 0 (0) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 2 (3) | 3 (5) | 2 (6) | 0 (0) | 3 (3)
Injection site reaction (General disorders) | 1 (2) | 6 (13) | 8 (32) | 0 (0) | 5 (20)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 2 (15) | 0 (0) | 2 (3)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (15) | 0 (0) | 6 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (5) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 2 (2) | 3 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 5 (6) | 4 (5) | 1 (1) | 5 (9)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal exfoliation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5) | 2 (2) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Myomectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days